CLINICAL TRIAL: NCT06959654
Title: The Diagnostic Value of Serum Oncostatin M and Galactin 3 as Biomarkers in Diagnosis of Ulcerative Colitis Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, manal mostafa kamel, Assistant lecture, Sohag University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: Soh-med-25-4-2MD
Record Dates: First submitted 2025-04-28; First posted 2025-05-06 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-04

CONDITIONS: Ulcerative Colitis Disease Patients and Normal Patients

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 :-normal healthy patients (Active Comparator): The study group will include 40 normal healthy subject.
  Interventions: Diagnostic Test: ELISA test
- Group2:-ulcerative colitis disease patients (Active Comparator): The study group will include 50 patients newly diagnosed with confirmed ulcerative colitis who divided into active and non active.
  Interventions: Diagnostic Test: ELISA test

INTERVENTIONS:
Diagnostic Test: ELISA test — ELISA test to evaulate serum oncostatin M and galactin 3 in two group of patientsL

SUMMARY:
Inflammatory bowel diseases (IBD)-Crohn's disease (CD), ulcerative colitis (UC) and inflammatory bowel disease unclassified (IBD-U)-are chronic inflammatory conditions that mainly affect the gastrointestinal tract but might also involve other organs, so they are considered systemic diseases. IBD is mainly diagnosed in young people, and is associated with significant morbidity and disability (Kaplan, 2015). Ulcerative colitis (UC) is an idiopathic, chronic inflammatory illness of the colon that is characterized by continous, diffuse mucosal inflammation (Ordás et al., 2012).

DETAILED DESCRIPTION:
Inflammatory bowel diseases (IBD)-Crohn's disease (CD), ulcerative colitis (UC) and inflammatory bowel disease unclassified (IBD-U)-are chronic inflammatory conditions that mainly affect the gastrointestinal tract but might also involve other organs, so they are considered systemic diseases. IBD is mainly diagnosed in young people, and is associated with significant morbidity and disability (Kaplan, 2015). Ulcerative colitis (UC) is an idiopathic, chronic inflammatory illness of the colon that is characterized by continous, diffuse mucosal inflammation (Ordás et al., 2012).

With 505 new cases per 100,000 people, Europe now has the highest prevalence of UC, followed by North America with 249 new cases per 100,000 people (Al-Fawzan et al., 2023), With an annual percentage rise of 4.3% (Kucharzik et al., 2020), it is becoming increasingly commonplace worldwide as more nations adopt Westernized lifestyles, leading to fast increases in incidence rates.

The aetiology involves interactions between the environment, immune system, gut microbiome and a genetic predisposition to disease (Kobayashi et al., 2020).

Ulcerative colitis presents with bloody diarrhea, frequency, abdominal pain, fatigue and faecal incontinence.

The pathogenesis of UC has not been elucidated yet, but it is supposed to be a consequence of unbalanced expression of molecules that have both anti- and pro-inflammatory properties (Ogino et al., 2021).

The inflammatory markers erythrocyte sedimentation rate (ESR), C-reactive protein (CRP), and fecal calprotectin (FC) have been studied to determine the type of ulcerative colitis (UC), its severity, prognosis, and responsiveness to treatment (Yuan et al., 2023).

Oncostatin M (OSM) is a proinflammatory cytokine belonging to the interleukin-6 family. OSM is produced mostly in hematopoietic tissues including T-lymphocytes, monocytes, macrophages, dendritic cells, neutrophils, eosinophils, and mast cells(West et al., 2018).

On the other hand, several pathological processes including arthritis, ossification, dermatitis, fibrosis, gingivitis, and carcinogenesis are found to have OSM mediation( Wolf et al., 2023).

One of the major pathological processes in which the involvement of OSM has been found critical is the inflammation of various parts including the joints, skin, lungs, and intestine(West et al., 2018).

The role of OSM in the pathogenesis of IBD was first described in a discovery of single nucleotide polymorphism in OSM receptors, OSM mediates its effects by binding to a glycoprotein called gp130 and this complex then activates the OSM receptor for signaling(Adrian-Segarra et al., 2018).

OSM is highly expressed in inflamed mucosa of IBD patients in comparison with normal individuals. Elevated OSM levels are also found in serum of IBD patients. Moreover, higher OSM levels are observed in first-degree relatives of multiple-affected families in comparison with normal families(Verstockt et al., 2019).

Galectins are a family of 15 (so far) mammalian galactoside-binding proteins that share a consensus amino acid sequence in their carbohydrate recognition domains (CRDs).

Based on their structural differences, galectin family members are classified into three subgroups of proto-, chimeric- and tandem-repeat-types. The prototype galectins include galectins-1, 2, 5, 7, 10, 11, 13, 14 and 15, each containing a single CRD in the polypeptide sequences and often identified as non-covalently linked homodimer.

The chimera-type galectin, which has only one member galectin-3, is composed of an unstructured non-lectin domain linked to a CRD and can form as multiple homotypic forms such as a pentamer. The tandem-repeat-type galectins include galectin-4, 6, 8, 9 and 12, each containing two different CRDs close to each end of the single polypeptide chain(Fred Brewer et al., 2002).

Interactions of galectins with galactose-terminated glycans on cell surface have also been implicated in the pathogenesis of IBD by induction of T cell apoptosis and NFkappa B signaling ( Paclik et al., 2008).

Level of serum galectin-3 was reported to be higher in IBD patients compared to healthy controls(Frol'ova et al., 2009). However, it is not known whether levels of any other galectin members are also altered in the circulation of IBD patients and whether serum galectins could be used as potential biomarkers for determining IBD and disease activity.

Rationale Endoscopic assessment is considered the gold standard for assessment of disease activity but repeated endoscopy is impractical, expensive and associated with poor patient acceptance and a potential for complications.

CRP is currently the most used non-invasive serum IBD biomarker in clinic. However, CRP determination limited by poor specificity and sensitivity as (i) CRP level isaltered in other acute inflammatory conditions in addition to CD and UC and (ii) up to 25% of patients, who have demonstrable disease activity determined by endoscopy have normal CRP values(Vermeire et al., 2004).

Fecal Calprotectin determination has far greater accuracy for detecting intestinal inflammation than CRP, but it requires collection of faecal sample which is cumbersome and has poor patient acceptability ( Marechal et al., 2017). Thus, there is a need for more accurate and non-invasive biomarkers for establishing disease activity in ulcerative colitis.

ELIGIBILITY:
Inclusion Criteria:

* Patients, both male and female, who are over the age of 18 and were identified as having ulcerative colitis based on histological, clinical, and endoscopic criteria.

Group I The study group will include 40 normal healthy subject. Group II The study group will include 50 patients newly diagnosed with confirmed ulcerative colitis who divided into active and non active.

Ulcerative colitis activity diagnosed by Simple Clinical Colitis Activity Index (SCCAI) is a diagnostic tool and questionnaire used to assess the severity of symptoms in people who suffer from ulcerative colitis(Walmsley et al.,1998). The calculated score ranges from 0 to20, where active disease is a score of 5 or higher. The score is determined by asking the person with colitis questions regarding:

Bowel frequency at day/night Urgency of defecation Blood in stool General health Extracolonic manifestations

Exclusion Criteria:

* Those with concomitant systemic inflammation as Rheumatoid arthritis(RA) and Bronchial asthma (BA), those with a history of malignancy, Also, patients who were discovered to have autoimmune disease or microscopic colitis and Crohn's disease, ulcerative colitis patients who are on treatment.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-05-15 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2028-05-15 (Estimated)

PRIMARY OUTCOMES:
Assessment of Serum value of oncosatin M and galactin 3 patients with ulcerative colitis | 1year
  - OSM and galactin 3 serum level measurement using the sandwich enzyme-linked immunosorbent test (ELISA), using a commercially available kit

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR